CLINICAL TRIAL: NCT00440037
Title: An Open Label Extension Study Evaluating the Safety and Efficacy of Long Term Dosing of AMG 531 in Thrombocytopenic Japanese Subjects With Immune (Idiopathic) Thrombocytopenic Purpura
Brief Title: Open Label Extension Study of AMG 531 in Japanese Subjects With ITP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060113; Japan CT Notification 18-1055 (Registry Identifier: Pharmaceuticals and Medical Devices Agency (PMDA))
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Keywords: AMG 531; ITP; Long term treatment; Japanese; Romiplostim
MeSH Terms: conditions — Purpura, Thrombocytopenic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 531 (Experimental)
  Interventions: Biological: AMG 531

INTERVENTIONS:
Biological: AMG 531 — AMG 531 will be administered by SC injection once per week from Week 1 (Day 1). The maximum permitted dose of AMG 531 is 10 μg/kg. AMG 531 will be supplied as a sterile, white, preservative-free, lyophilized powder in 5 mL glass vials containing 0.6 mg of protein per vial, and a protein concentration of 0.5 mg/mL when reconstituted with 1.2 mL of sterile water for injection.
  Other Names: Romiplostim

SUMMARY:
The purpose of this study is to assess the safety and efficacy of long term dosing of AMG 531 in thrombocytopenic Japanese subjects with ITP.

It is anticipated that AMG 531 will be a safe and well tolerated in long term treatment and that AMG 531 will effectively raise and maintain platelet counts to a desired therapeutic range, when individual dose adjustments based on platelet counts are permitted.

This study is available to subjects who have completed any previous AMG 531 ITP study in Japan and meet the eligibility criteria of this study.

DETAILED DESCRIPTION:
Romiplostim was administered by subcutaneous (SC) injection once per week. If subjects entered the extension study within 12 weeks from the last investigational product administration in the previous study and had shown an increase in platelet counts ≥ 20 x 109/L from baseline at least once during the 13-week treatment period (excluding 4 weeks after receiving rescue medication), they were treated with romiplostim at the same weekly dose (last dose on study) received in the previous study. Otherwise, subjects were treated with romiplostim at a starting dose of 3 μg/kg. Dose adjustment based on platelet counts was allowed throughout the treatment period to allow subjects to maintain platelet counts in the target range of ≥ 50 to ≤ 200 x 109/L, up to a maximum permitted dose of 10 μg/kg.

ELIGIBILITY:
Inclusion Criteria

* Subjects must have previously completed an AMG 531 ITP study in Japan.
* Platelet count taken at the screening visit must be < 50 x 109/L.
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria

* Any significant change in medical history since completion of the previous AMG 531 ITP study including bone marrow stem cell disorders or new active malignancies
* known positive result from a test for neutralizing antibodies to AMG 531 in the previous AMG 531 ITP study
* Currently receiving any treatment for ITP except oral corticosteroids, azathioprine and/or danazol administered at a constant dose and schedule from at least 4 weeks prior to the screening visit
* received intravenous immunoglobulin, anti-D immunoglobulin, or any drug administered to increase platelet counts (eg, immunosuppressants etc) within 1 week before the screening visit
* received anti-malignancy agents (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, Interferon-alfa etc) within 4 weeks before the screening visit
* received any monoclonal antibody drugs (eg, rituximab etc) within 8 weeks before the screening visit
* Less than 4 weeks since receipt of any therapeutic drug or device that is not Ministry of Health, Labor and Welfare (MHLW) approved for any indication before the screening visit (excluding AMG 531)
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator
* known severe drug hypersensitivity
* Concerns for subject's compliance with the protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-11; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- Japan (11):
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Isehara-shi, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Suita, Osaka
  - Research Site, Chūō
  - Research Site, Hirakata
  - Research Site, Hiroshima
  - Research Site, Kumamoto
  - Research Site, Moriguchi
  - Research Site, Tokyo

REFERENCES:
- [Derived] Arranz R, Garcia-Noblejas A, Grande C, Cannata-Ortiz J, Sanchez JJ, Garcia-Marco JA, Alaez C, Perez-Calvo J, Martinez-Sanchez P, Sanchez-Gonzalez B, Canales MA, Conde E, Martin A, Arranz E, Terol MJ, Salar A, Caballero D. First-line treatment with rituximab-hyperCVAD alternating with rituximab-methotrexate-cytarabine and followed by consolidation with 90Y-ibritumomab-tiuxetan in patients with mantle cell lymphoma. Results of a multicenter, phase 2 pilot trial from the GELTAMO group. Haematologica. 2013 Oct;98(10):1563-70. doi: 10.3324/haematol.2013.088377. Epub 2013 Jun 10. PMID 23753021
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had completed any previous romiplostim ITP study in Japan (Studies 20050162/NCT00305435 or 20060216/NCT00603642) were eligible to screen for this study. The study began in October 2006 and continued until romiplostim was commercially available in Japan.
Groups:
- AMG 531: AMG531 was administered by SC injection once per week from Week 1 (Day 1). The maximum permitted dose of AMG531 was 10 μg/kg.
Period: Overall Study
Arm/Group | AMG 531
Started | 44
Completed | 35
Not Completed | 9
Not completed — Withdrawal by Subject | 6
Not completed — Administrative decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | AMG 531
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 44
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events Including Clinically Significant Changes in Laboratory Values.
Description: Subjects who reported at least 1 adverse event after beginning treatment with romiplostim in this study
Time Frame: Through study completion, the median treatment duration (time between first dose and last dose) was 146.0 weeks (range: 12 to 243 weeks)
Population: Subjects in Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AMG 531
Number analyzed (Participants) | 44
percentage of participants | 100

2. Secondary Outcome: Incidence of Anti AMG 531 Antibody Formation
Description: Subjects with positive anti-AMG 531 antibodies (either to the peptide portion of AMG 531 or to the intact molecule) and antibodies that cross-react with endogenous thrombopoietin (TPO)
Time Frame: as for outcome 1
Population: Subjects with at least 1 immunoassay available
Measure: Number; unit: percentage of participants
Arm/Group | AMG 531
Number analyzed (Participants) | 44
percentage of participants
  Positive for romiplostim-neutralizing antibodies | 0
  Positive for TPO-neutralizing antibodies | 0

3. Secondary Outcome: Incidence of Platelet Response (Platelet Response is Defined as a Doubling of Baseline Platelet Counts and More Than 50 x 10^9/L; Baseline Platelet Counts is That Obtained in the Previous Study)
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 531
Number analyzed (Participants) | 44
percentage of participants | 95.5 [84.5 to 99.4]

4. Secondary Outcome: Percentage of Subjects Able to Reduce or Discontinue Their Concurrent ITP Therapies (for Subjects That Are Receiving Oral Corticosteroids at a Constant Dose and Schedule at the Screening Visit)
Time Frame: as for outcome 1
Population: Subjects who were receiving concurrent ITP therapy at baseline
Measure: Number; unit: percentage of participants
Arm/Group | AMG 531
Number analyzed (Participants) | 25
percentage of participants | 100

5. Secondary Outcome: Change From Baseline in Patient-reported Outcome (PRO) Endpoints at Each Time Point (Baseline PRO is Obtained at Day 1 Predose)
Description: Short Form 36 (SF-36): The SF-36 has 36 questions with 8 domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health. In addition to deriving a score for each of the domains, the SF-36 generates 2 summary scores: a physical component summary (PCS) and a mental component summary (MCS). These 8 domains and 2 summary scores are scored from 0 to 100, with higher scores indicating better health status. The official version in Japanese was used in this study.
  Euroqol-5 Dimensions (EQ-5D): The EQ-5D is a patient-completed, multidimensional measure of HRQOL. EQ-5D index values range from -0.59 to 1.00. The EQ-5D visual analogue scale (VAS) records the respondents' self-rated health status on a vertical graduated (0 to 100) visual analogue scale. Higher EQ-5D Index and VAS scores represent better health status. The official version in Japanese was used in this study.
Time Frame: By Week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AMG 531
Number analyzed (Participants) | 44
score on a scale
  Change in EQ-5D Index score at Week 48 | 0.02 (0.12)
  Change in EQ-5D VAS score at Week 48 | 6.13 (16.48)
  Change in SF-36 physical functioning at Week 48 | 0.68 (7.19)
  Change in SF-36 role physical at Week 48 | 2.30 (10.43)
  Change in SF-36 bodily pain at Week 48 | -0.87 (13.42)
  Change in SF-36 General Health Perception at W48 | 1.30 (5.14)
  Change in SF-36 Vitality at Week 48 | 1.12 (8.42)
  Change in SF-36 Social Functioning at Week 48 | 1.22 (8.56)
  Change in SF-36 Role Emotional at Week 48 | 1.84 (12.82)
  Change in SF-36 Mental Health at Week 48 | -1.42 (9.04)
  Change in SF-36 Physical Component at Week 48 | 1.13 (6.85)
  Change in SF-36 Mental Component at Week 48 | 0.33 (9.19)

ADVERSE EVENTS:
Time Frame: The duration of treatment in this study ranged from 12 to 243 weeks; the median (Q1, Q3) duration of treatment in this study was 146.0 (119.5, 166.0) weeks.
Arm/Group | AMG 531
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 12/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 531 (N=44)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1
Feeling Abnormal (General disorders) | 1
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 1
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Grand Mal Convulsion (Nervous system disorders) | 1
Intracranial Aneurysm (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 531 (N=44)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Vertigo (Ear and labyrinth disorders) | 8
Conjunctival Haemorrhage (Eye disorders) | 3
Conjunctivitis (Eye disorders) | 4
Abdominal Discomfort (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 8
Colonic Polyp (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Dental Caries (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 7
Gastritis (Gastrointestinal disorders) | 4
Gingivitis (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Malaise (General disorders) | 8
Oedema Peripheral (General disorders) | 3
Pyrexia (General disorders) | 4
Hepatic Function Abnormal (Hepatobiliary disorders) | 4
Bronchitis (Infections and infestations) | 3
Cystitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 35
Pharyngitis (Infections and infestations) | 5
Arthropod Sting (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 9
Excoriation (Injury, poisoning and procedural complications) | 6
Laceration (Injury, poisoning and procedural complications) | 3
Thermal Burn (Injury, poisoning and procedural complications) | 4
Wound (Injury, poisoning and procedural complications) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 12
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8
Headache (Nervous system disorders) | 19
Hypoaesthesia (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 7
Eczema (Skin and subcutaneous tissue disorders) | 7
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes